CLINICAL TRIAL: NCT00683241
Title: A Phase I Clinical Trial of Autologous Dendritic Cell Vaccine Leaded With Autologous Tumor Cell Lysate for Recurrent Ovarian or Primary Peritoneal Cancer
Brief Title: A Phase I Clinical Trial of Autologous Dendritic Cell Vaccine for Recurrent Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Northwest Biotherapeutics (Industry); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 11807
Record Dates: First submitted 2008-05-19; First posted 2008-05-23 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Ovarian Cancer; Peritoneal Cancer
Keywords: Vaccine; Ovarian; Peritoneal
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Subjects with stage II to IV recurrent epithelial ovarian carcinoma or recurrent primary peritoneal cancer, from whom solid tumor, ascites or pleural effusion will be harvested and available and sufficient for lysate preparation; and whose largest tumor nodule is ≤ 2.5 cm. Subjects may have undergone chemotherapy or other therapy following tumor harvesting and prior to enrollment (apheresis).
  Interventions: Biological: DCVac-L

INTERVENTIONS:
Biological: DCVac-L — Subjects will receive three doses of intradermal vaccination with ~5-10 x 106 dendritic cells (DCVax-L) on days 0, 14 and 28

SUMMARY:
This study is open to women with recurrent epithelial ovarian carcinoma or primary peritoneal cancer. Subjects will be asked to donate either a piece of their tumor or malignant effusion in order to make the first part of the vaccine or lysate. If enough of the lystate had been collected to make the first part of the vaccine, then subjects may enroll in the study as long as they meet the rest of the entry criteria.

After is determined that a subject is eligible to enroll into the study, you will have to donate some blood in order to make the second part of the vaccine. After this, the blood and vaccine are mixed together to make the vaccine called DCVax-L. You will be given two dose of a drug called Avastin every other week (Avastin will be given through your vein) and a oral chemotherapy called Cytoxan. One week after your last dose of oral Cytoxan, you will receive 3 vaccines given every other week for the next month. After the first two doses of vaccine, you will also receive more Avastin. During the study you will be seeing your study team to have physical exams, blood drawn in order to monitor your health and have blood drawn for research. The study team will contact you for the next 5 years in order to determine how you are doing.

DETAILED DESCRIPTION:
Subjects with recurrent epithelial ovarian carcinoma or recurrent primary peritoneal cancer, for whom autologous tumor or malignant effusion has been harvested and is available for lysate preparation, are eligible, provided all other eligibility criteria are fulfilled. Harvested tumor or malignant effusion will be shipped to Cognate BioServices (Sunnyvale, CA) for preparation of lysate. If sufficient amount of lysate for vaccine can be generated, subjects will be enrolled to the study.

Subjects will undergo apheresis on day -35 to -29 to harvest peripheral blood mononuclear cells (PBMC). The apheresis product will be shipped to Cognate BioServices, where DC will be prepared and pulsed with autologous lysate according to proprietary technology. Following apheresis, subjects will receive two cycles of biological antiangiogenesis/immunomodulatory therapy comprising intravenous bevacizumab at 10 mg/kg on day -28 and -14, which may be followed by 7 days of oral metronomic cyclophosphamide at 50 mg daily (days -28 to -21, and -14 to -7, respectively). Subjects will receive three doses of intradermal vaccination with ~5-10 x 106 dendritic cells (DCVax-L) on days 0, 14 and 28. Subjects will also receive intravenous bevacizumab at 10 mg/kg concurrently with intradermal DCVax-L on day 0 and 14, which may be followed by oral cyclophosphamide at 50 mg for 7 days (days 0 to 7, and 14 to 21, respectively). The last DCVax-L (day 28) may be followed by oral cyclophosphamide at 50 mg daily x 7 days (days 28 to 35), but no bevacizumab will be given on day 28. Prevnar, an FDA approved seven-valent vaccine against Pneumococcus pneumoniae, will be given intramuscularly on day 0 as positive control of immune responsiveness. Two weeks following third vaccine dose (day 42), patients will undergo immune assessment.

Subjects will be contacted every 6 months for 5 years and then annually for survival. Subject will have the option of enrolling in other combinatorial immunotherapy trials when these are available, if they satisfy enrollment criteria. Subjects will have the option of continuing vaccination every two months till exhaustion of DCVax-L or disease progression, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent stage II to IV ovarian carcinoma or primary peritoneal carcinoma.
* Subjects with prior secondary cytoreductive surgery or aspiration of malignant effusion yielding tumor for lysate preparation.
* Subjects must have sufficient lysate for DCVax-L preparation (> 10 mg of pure protein lysate from tumor, ascites or malignant pleural effusion cell preparation).
* largest tumor nodule ≤ 2.5 cm
* Patients who have achieved complete response following surgery and chemotherapy are still eligible for vaccine.
* may be platinum-sensitive or platinum-resistant
* may have received chemotherapy or other therapy after harvest of tumor
* must have recovered from toxicities of prior chemotherapy or other therapy.
* completed all parenteral investigational therapy 14 days and have completed all oral investigational therapy 7 days prior to enrollment
* must have completed all hormonal therapy 7 days prior to enrollment.
* must have recovered from toxicities of radiation therapy (to grade 2 or less).
* at least 4 weeks postoperative recovery
* coagulation studies w/i normal limits
* ECOG > 2
* Life expectancy of > 4 months.
* must understand and sign the study specific informed consent.

Exclusion Criteria:

* not enough lysate for vaccine preparation
* known brain metastases
* any of the following positive tests at the screening visit: (HTLV-1/2 ; Hepatitis B, HIV, Hepatitis C, Anti-Yo(cdr2) antibody present in serum
* on corticosteroids
* prior IV Cytoxan at maximally tolerated dose
* serum creatinine > 2.2 mg/dl or BUN > 40 mg/dl
* proteinuria > 3.5gm over 24 hrs
* serum total bilirubin > 2.0 and/or serum transaminases > 3X the upper limits of normal
* Platelets < 100,000/ mm3 ; WBC < 3,000/mm3 ; Absolute Neutrophil Count (ANC) < 1,500/mm3 ; Absolute lymphocyte count < 1000/ mm3 ; Hematocrit < 30%
* acute infection that requires specific therapy
* serious, non-healing wound, ulcer, or bone fracture
* active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6 months of the first date of treatment on this study.
* clinically significant cardiovascular disease; this includes: (Uncontrolled hypertension ; Myocardial infarction or unstable angina within 6 months prior to registration ; New York Heart Association (NYHA) Grade II or greater congestive heart failure ; Serious cardiac arrhythmia requiring medication ; Grade II or greater peripheral vascular disease.
* clinically significant peripheral artery disease, e.g., those with claudication, within 6 months.
* clinical symptoms or signs of partial or complete gastrointestinal obstruction or who require parenteral hydration and/or nutrition.
* any underlying conditions which would contraindicate therapy with study treatment (or allergies to reagents used in this study). Subjects with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
* organ allografts.
* known autoimmune/collagen vascular disorder.
* on any medications that might affect immune function. Additionally, H2 antagonists are excluded as are all antihistamines five days before and five days after each injection of study drug. NSAIDS including COX-2 inhibitors, acetaminophen or aspirin are exceptions.
* pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and safety of administering DCVax-L intradermally combined with intravenous bevacizumab and oral metronomic cyclophosphamide in patients with recurrent ovarian or primary peritoneal cancer. | 2 years

SECONDARY OUTCOMES:
To assess the immunogenicity of DCVax-L administered intradermally in patients with recurrent ovarian or recurrent primary peritoneal cancer, combined with intravenous bevacizumab and oral metronomic cyclophosphamide. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: George Coukos, M.D., Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Gynecologic Oncology @ University of Pennsylvania — http://pennhealth.com/WagForm/MainPage.aspx?config=provider&P=LP&ID=279